CLINICAL TRIAL: NCT02640794
Title: Aspirin Versus Aspirin + ClopidogRel as Antithrombotic Treatment Following Transcatheter Aortic Valve Implantation With the Edwards Valve. A Randomized Study (the ARTE Trial)
Brief Title: Aspirin Versus Aspirin+Clopidogrel as Antithrombotic Treatment Following TAVI
Acronym: ARTE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Responsible Party: Principal Investigator, Josep Rodes-Cabau, MD, Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec
Organization: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ARTE2
Record Dates: First submitted 2015-12-23; First posted 2015-12-29 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Aortic Valve Disease; Myocardial Infarction; Stroke; Bleeding
Keywords: Transcatheter aortic valve implantation; Antithrombotic treatment; Clopidogrel; Aspirin/acetylsalicylic acid; Myocardial Infarction; Ischemic stroke; Major bleeding
MeSH Terms: conditions — Aortic Valve Disease; Myocardial Infarction; Stroke; Hemorrhage; Ischemic Stroke | interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspirin +clopidogrel (Active Comparator): Patients would be randomized within the month prior to the TAVI procedure to receive aspirin/acetylsalicylic acid (80-325 mg/d) + clopidogrel (75 mg/d)
  Interventions: Drug: Clopidogrel; Drug: Aspirin
- Aspirin (Active Comparator): Patients will be randomized within the month prior to the TAVI procedure to receive aspirin/acetylsalicylic acid (80-325 mg/d)
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel therapy will start within 24 hrs before the TAVI procedure in cases where a transfemoral approach is used and within 24 hrs after the TAVI procedure in cases where a transapical approach is used. The initial dose of clopidogrel will be of 300 mg followed by 75 mg/die. The duration of clopidogrel treatment will be of 3 months.
  Other Names: Plavix
  Arms: Aspirin +clopidogrel
Drug: Aspirin — Aspirin/acetylsalicylic acid (80-325 mg/d). Aspirin/acetylsalicylic acid therapy will start at least 24 hrs before the TAVI procedure and continued for at least 6 months.
  Other Names: Acetylsalicylic acid

SUMMARY:
The purpose of this study is to compare aspirin/acetylsalicylic acid+ clopidogrel with aspirin/acetylsalicylic acid alone as antithrombotic treatment following TAVI for the prevention of major ischemic events (MI, ischemic stroke) or death without increasing the risk of major bleeding events.

DETAILED DESCRIPTION:
Transcatheter aortic valve implantation (TAVI) has emerged as an alternative to standard aortic valve replacement for the treatment of patients considered to be at very high or prohibitive surgical risk. Nowadays the procedure is associated with a very high success rate (>95%) but major peri-procedural ischemic complications such as myocardial infarction (MI) or ischemic stroke occur in about 2% (0% to 17%) and 3% (2% to 7%) of the cases, respectively. The recently published PARTNER trial showed a stroke rate as high as 6.5% within the 30 days following TAVI, with most (77%) of these events diagnosed as major strokes. In order to avoid such ischemic complications full dose anticoagulation (usually intravenous heparin) is administered during the TAVI procedure, whereas aspirin (long-term) + clopidogrel (1 to 6 months) have been the recommended antithrombotic treatment following the procedure. However, this antithrombotic regime has been recommended on an empirical basis, and no studies have as yet shown the efficacy of aspirin + clopidogrel vs. aspirin alone or no antithrombotic treatment in preventing ischemic events following TAVI procedures. Also, patients undergoing TAVI nowadays are usually octogenarians and very frequently exhibit comorbidities such as hypertension, abnormal renal function or prior cerebrovascular disease, which significantly increase the risk of major bleeding. Indeed, TAVI procedures can also be associated with major vascular complications which in turn can complicate with life-threatening or major bleeding. It is well know that clopidogrel on top of aspirin is associated with a higher rate of major bleeding complications, especially in elderly patients. It would therefore be of major clinical relevance to determine the risk/benefit ratio of using a dual antithrombotic therapy following TAVI procedures in order to recommend the most appropriate antithrombotic treatment in this high-risk population. The ARTE trial is a multicenter randomized study to evaluate the efficacy and safety of aspirin/acetylsalicylic acid versus aspirin/acetylsalicylic acid+ clopidogrel as antithrombotic treatment after TAVI.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a TAVI procedure with the Edwards valve.

Exclusion Criteria:

* Need for chronic anticoagulation treatment
* Major bleeding within the 3 months prior to the TAVI procedure
* Prior intracranial bleeding
* Drug-eluting stent implantation within the year prior to the TAVI procedure
* Allergy to clopidogrel and/or aspirin/acetylsalicylic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Incidence of death, MI, ischemic stroke/Transient ischemic attack (TIA) or life threatening/major bleeding at 3-month follow-up. | 3-month follow-up
  The composite endpoint of incidence of death, MI, ischemic stroke/Transient ischemic attack (TIA) or life life threatening/major bleeding at 3-month follow-up will be analyzed

SECONDARY OUTCOMES:
Incidence of death, MI, ischemic stroke/TIA or life threatening/major bleeding at 30 days | 30 days
  The composite endpoint of Incidence of death, MI, ischemic stroke/TIA or life threatening/major bleeding at 30 days will be analyzed
Incidence of death, MI, ischemic stroke/TIA or life threatening/major bleeding at at 12-month follow-up | 12-month follow-up
  The composite endpoint of Incidence of death, MI, ischemic stroke/TIA or life threatening/major bleeding at at 12-month follow-up will be analyzed.
Incidence of MI or ischemic stroke at 30 days and at 12-month follow-up | 12-month follow-up
  The composite endpoint of incidence of MI or ischemic stroke at 30 days and at 12-month follow-up will be analyzed
Cardiovascular death at 30 days and at 12-month follow-up | 30 days and at 12-month follow-up
  The incidence of cardiovascular death at 30 days and at 12-month follow-up will be analyzed
Cost-effectiveness of clopidogrel on top of aspirin/acetylsalicylic acid following TAVI | 30 days and at 12-month follow-up
  Cost-effectiveness of clopidogrel on top of aspirin/acetylsalicylic acid following TAVI will be analyzed
Rate of minor bleeding at 30 days and at 12-month follow-up | 30 days and at 12-month follow-up
  Rate of minor bleeding at 30 days and at 12-month follow-up will be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Josep Rodes, MD, Principal Investigator — Fondation IUCPQ
Locations (4):
- Canada (2):
  - St Michael's Hospital, Toronto, Ontario
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec
- Hospital San Borja Arriaran, Santiago, Chile
- Hospital Vall d'Hebron de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rodes-Cabau J. [Progress in transcatheter aortic valve implantation]. Rev Esp Cardiol. 2010 Apr;63(4):439-50. Spanish. PMID 20334810
- [Result] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243
- [Result] Thomas M, Schymik G, Walther T, Himbert D, Lefevre T, Treede H, Eggebrecht H, Rubino P, Michev I, Lange R, Anderson WN, Wendler O. Thirty-day results of the SAPIEN aortic Bioprosthesis European Outcome (SOURCE) Registry: A European registry of transcatheter aortic valve implantation using the Edwards SAPIEN valve. Circulation. 2010 Jul 6;122(1):62-9. doi: 10.1161/CIRCULATIONAHA.109.907402. Epub 2010 Jun 21. PMID 20566953
- [Result] Rodes-Cabau J, Webb JG, Cheung A, Ye J, Dumont E, Feindel CM, Osten M, Natarajan MK, Velianou JL, Martucci G, DeVarennes B, Chisholm R, Peterson MD, Lichtenstein SV, Nietlispach F, Doyle D, DeLarochelliere R, Teoh K, Chu V, Dancea A, Lachapelle K, Cheema A, Latter D, Horlick E. Transcatheter aortic valve implantation for the treatment of severe symptomatic aortic stenosis in patients at very high or prohibitive surgical risk: acute and late outcomes of the multicenter Canadian experience. J Am Coll Cardiol. 2010 Mar 16;55(11):1080-90. doi: 10.1016/j.jacc.2009.12.014. Epub 2010 Jan 22. PMID 20096533
- [Result] Gurvitch R, Wood DA, Tay EL, Leipsic J, Ye J, Lichtenstein SV, Thompson CR, Carere RG, Wijesinghe N, Nietlispach F, Boone RH, Lauck S, Cheung A, Webb JG. Transcatheter aortic valve implantation: durability of clinical and hemodynamic outcomes beyond 3 years in a large patient cohort. Circulation. 2010 Sep 28;122(13):1319-27. doi: 10.1161/CIRCULATIONAHA.110.948877. Epub 2010 Sep 13. PMID 20837893
- [Result] Lip GY, Nieuwlaat R, Pisters R, Lane DA, Crijns HJ. Refining clinical risk stratification for predicting stroke and thromboembolism in atrial fibrillation using a novel risk factor-based approach: the euro heart survey on atrial fibrillation. Chest. 2010 Feb;137(2):263-72. doi: 10.1378/chest.09-1584. Epub 2009 Sep 17. PMID 19762550
- [Result] Shehab N, Sperling LS, Kegler SR, Budnitz DS. National estimates of emergency department visits for hemorrhage-related adverse events from clopidogrel plus aspirin and from warfarin. Arch Intern Med. 2010 Nov 22;170(21):1926-33. doi: 10.1001/archinternmed.2010.407. PMID 21098354
- [Result] ACTIVE Investigators; Connolly SJ, Pogue J, Hart RG, Hohnloser SH, Pfeffer M, Chrolavicius S, Yusuf S. Effect of clopidogrel added to aspirin in patients with atrial fibrillation. N Engl J Med. 2009 May 14;360(20):2066-78. doi: 10.1056/NEJMoa0901301. Epub 2009 Mar 31. PMID 19336502
- [Result] Hansen ML, Sorensen R, Clausen MT, Fog-Petersen ML, Raunso J, Gadsboll N, Gislason GH, Folke F, Andersen SS, Schramm TK, Abildstrom SZ, Poulsen HE, Kober L, Torp-Pedersen C. Risk of bleeding with single, dual, or triple therapy with warfarin, aspirin, and clopidogrel in patients with atrial fibrillation. Arch Intern Med. 2010 Sep 13;170(16):1433-41. doi: 10.1001/archinternmed.2010.271. PMID 20837828
- [Result] Delaney JA, Opatrny L, Brophy JM, Suissa S. Drug drug interactions between antithrombotic medications and the risk of gastrointestinal bleeding. CMAJ. 2007 Aug 14;177(4):347-51. doi: 10.1503/cmaj.070186. PMID 17698822
- [Result] Leon MB, Piazza N, Nikolsky E, Blackstone EH, Cutlip DE, Kappetein AP, Krucoff MW, Mack M, Mehran R, Miller C, Morel MA, Petersen J, Popma JJ, Takkenberg JJ, Vahanian A, van Es GA, Vranckx P, Webb JG, Windecker S, Serruys PW. Standardized endpoint definitions for transcatheter aortic valve implantation clinical trials: a consensus report from the Valve Academic Research Consortium. Eur Heart J. 2011 Jan;32(2):205-17. doi: 10.1093/eurheartj/ehq406. Epub 2011 Jan 6. PMID 21216739
- [Derived] Rodes-Cabau J, Masson JB, Welsh RC, Garcia Del Blanco B, Pelletier M, Webb JG, Al-Qoofi F, Genereux P, Maluenda G, Thoenes M, Paradis JM, Chamandi C, Serra V, Dumont E, Cote M. Aspirin Versus Aspirin Plus Clopidogrel as Antithrombotic Treatment Following Transcatheter Aortic Valve Replacement With a Balloon-Expandable Valve: The ARTE (Aspirin Versus Aspirin + Clopidogrel Following Transcatheter Aortic Valve Implantation) Randomized Clinical Trial. JACC Cardiovasc Interv. 2017 Jul 10;10(13):1357-1365. doi: 10.1016/j.jcin.2017.04.014. Epub 2017 May 17. PMID 28527771